CLINICAL TRIAL: NCT00138008
Title: Randomized Controlled Trial to Evaluate Radiotherapy Followed by Endocrine Therapy vs. Endocrine Therapy Alone for PSA Failure After Radical Prostatectomy (JCOG0401)
Brief Title: Trial to Evaluate Radiotherapy Followed by Endocrine Therapy Vs Endocrine Therapy Alone for PSA Failure After Radical Prostatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0401; C000000026 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radical prostatectomy; PSA failure; RCT; radiation; endocrinotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Drug: endocrine therapy
  Interventions: Drug: endocrine therapy
- 2 (Experimental): Procedure/Surgery: radiotherapy
  Interventions: Procedure: radiotherapy

INTERVENTIONS:
Drug: endocrine therapy — Drug: endocrine therapy
  Arms: 1
Procedure: radiotherapy — Procedure/Surgery: radiotherapy
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate radiotherapy followed by endocrine therapy in comparison with endocrine therapy alone for PSA failure after radical prostatectomy.

DETAILED DESCRIPTION:
A randomized controlled trial is conducted in Japan to evaluate radiotherapy followed by endocrine therapy for PSA failure after radical prostatectomy. Patients who have PSA failure after radical prostatectomy under a diagnosis of localized prostate cancer (T1-2 N0M0) are randomized into treatment group of either radiotherapy followed by endocrine therapy or endocrine therapy alone. Urologic Oncology Study Group (UOSG) in the JCOG composed of 36 specialized institutions will recruit 200 patients. The primary endpoint is time to treatment failure (TTF) of bicalutamide and secondary endpoints are TTF of protocol treatment, progression free survival, overall survival, adverse events and quality of life (QOL). The Clinical Trial Review Committee of the Japan Clinical Oncology Group (JCOG) approved the protocol on April 13, 2004, and the study was activated on May 17, 2004.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of localized prostate cancer (clinical stage T1-2N0M0) which is treated by radical prostatectomy
* Pathological stage: pT0/2/3 and pN0/x
* Serum level of PSA once reached < 0.1 ng/ml after radical prostatectomy and then increased 0.4 ng/ml
* Serum level of PSA 1.0 ng/ml at entry
* No clinical recurrence based on abdominal and pelvic computed tomography, and a bone scan
* No history of chemotherapy or radiation therapy or endocrine therapy for any cancer
* Ages 20 to 79 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* No blood transfusion within 28 days of entry
* Sufficient organ function within 28 days of entry
* Provided written informed consent

Exclusion Criteria:

* Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ
* Mental disease or mental symptoms which would affect participant's decision to participate
* Continuous medication with steroids (exclude external use of steroids for skin)
* Ischemic heart disease or arrhythmia which needs medical treatment
* Poorly controlled hypertension
* Poorly controlled diabetes mellitus
* History of cerebral infarction or myocardial infarction within 6 months
* Liver cirrhosis
* Interstitial pneumonia which requires ventilation assistance, oxygen inhalation, steroids, or diuretic medicine

Ages: 20 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
time to treatment failure (TTF) of bicalutamide | time to treatment failure (TTF) of bicalutamide

SECONDARY OUTCOMES:
TTF of protocol treatment | TTF of protocol treatment
clinical progression free survival | time to clinical progression
overall survival | overall
adverse events | overall
patient-reported quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Seiji Naito, MD, Ph.D., Study Chair — Graduate School of Medical Science, Kyushu University
Locations (34):
- Japan (34):
  - Nagoya University School of Medicine, Nagoya,Showa-ku,Tsurumai-cho,65, Aichi-ken
  - Akita University School of Medicine, Akita,Hondo,1-1-1, Akita
  - Chiba University, Graduate School of Medicine, Chiba,Chuo-ku,Inohana,1-8-1, Chiba
  - Chiba Cancer Center Hospital, Chiba,Chuo-ku,Nitona-cho,666-2, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Graduate School of Medical Science, Kyushu University, Fukuoka, Higashi-ku,Maidashi,3-1-1, Fukuoka
  - Kurume University School of Medicine, Kurume,Asahi-machi,67, Fukuoka
  - Gunma University, Maebashi,Showa,3-39-15, Gunma
  - Hokkaido University Hospital, North-14 West-5 Kita-ku,Sapporo, Hokkaido
  - Sapporo Medical University, S-1,W-16,Chuo-ku,Sapporo, Hokkaido
  - Kobe University Graduate School of Medicine, Kobe,Chuo-ku,Kusunoki-cho,7-5-2, Hyōgo
  - Institute of Clinical Medicine,Tsukuba University Hospital, Tsukuba,Tennodai,1-1-1, Ibaraki
  - Faculty of Medicine, Kagawa University, Kita,Miki-cho,Ikenobe,1750-1, Kagawa-ken
  - Kagoshima University,Faculty of Medicine, Kagoshima,Sakuragaoka,8-35-1, Kagoshima-ken
  - Kitasato University School of Medicine, Sagamihara,Kitasato,1-15-1, Kanagawa
  - Kyoto University Hospital, Kyoto,Sakyo-ku,Syogoinkawara,54, Kyoto
  - Mie University School of Medicine, Tsu,Edobashi,2-174, Mie-ken
  - Miyagi Cancer Center, Natori,Medeshima-Shiode,Nodayama,47-1, Miyagi
  - Tohoku University Hospital, Sendai,Aoba-ku,Seiryo-machi,1-1, Miyagi
  - Sinshu University, Matsumoto,Asahi,3-1-1, Nagano
  - Nara Medical University, Kashihara,Shijo-cho,840, Nara
  - Niigata University Medical and Dental Hospital, Niigata,Asahimachi-dori,1-754, Niigata
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Kurashiki Central Hospital, Kurashiki,Miwa,1-1-1, Okayama-ken
  - Okayama University Hospital, Okayama,Shikata-cho,2-5-1, Okayama-ken
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Shimane University Faculty of Medicine, Izumo,Enya-cho,89-1, Shimane
  - Hamamatsu University School of Medicine, Hamamatsu,Handayama,1-20-1, Shizuoka
  - Sizuoka Cancer Center, Sunto-gun,Nagaizumi-cho,Shimonagakubo,1007, Shizuoka
  - Tochigi Cancer Center, Utsunomiya,Yohnan,4-9-13, Tochigi
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - Jikei University Hospital, Minato-ku,Nishishinbashi,3-25-8, Tokyo
  - Keio University Hospital, Shinjuku-ku,Shinanomachi,35, Tokyo
  - University of Yamanashi Faculty of Medicine, Nakakoma,Tamaho,Shimokato,1110, Yamanashi

REFERENCES:
- See also: Related Info — http://www.jcog.jp/